CLINICAL TRIAL: NCT04150458
Title: Performance of 18F-Fluorocholine Positron Emission Tomography With Computed Tomography in Patients With 18F-Fluorocholine-avid Lesions: A Basket Trial
Brief Title: Fluorocholine PET/CT Basket Trial
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FCH Basket
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fluorocholine PET/CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorocholine PET/CT (Experimental): The sole study-specific procedure is a single 18F-fluorocholine positron emission tomography / computed tomography (PET/CT). Subjects will receive 9 mCi 18F-fluorocholine IV, 5 to 120 minutes prior to PET/CT. 18F-fluorocholine PET/CT studies will be performed on hybrid PET/CT scanners which combine a dedicated, full-ring PET scanner with a multi-slice spiral CT scanner.
  Interventions: Drug: 18F-fluorocholine PET/CT.

INTERVENTIONS:
Drug: 18F-fluorocholine PET/CT. — 18F-fluorocholine positron emission tomography / computed tomography
  Other Names: FCH PET/CT; F-choline PET/CT

SUMMARY:
This is a single-arm, open-label, phase III trial in up to 2000 patients with known or suspected benign or malignant tumors which are known or suspected to be 18F-fluorocholine-avid.

Patients will receive regular standard clinical care. The only study-specific procedure will be the administration of 18F-fluorocholine followed by a PET/CT scan.

Diagnostic accuracy of 18F-fluorocholine PET/CT will be captured versus a composite clinical, radiological and histopathological standard of truth at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Under referring physician's care
* Able to understand and provide written informed consent
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine (or prone) for up to 30 minutes and tolerating intravenous cannulation for injection
* Known or suspected benign or malignant tumor which is known or suspected to be 18F-fluorocholine-avid as per current medical literature

Exclusion Criteria:

* Medically unstable (e.g. acute cardiac or respiratory distress or hypotensive)
* Exceeding the safe weight limit of the PET/CT bed (usually approximately 400 lbs.) or cannot fit through the PET/CT bore (usually approximately 70 cm diameter)
* Unmanageable claustrophobia

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Fluorocholine PET/CT | 1 day
  Sensitivity, specificity, positive predictive and negative predictive values of 18F-fluorocholine PET/CT in the detection of tumor lesions as compared to a composite truth standard.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events following Fluorocholine PET/CT | 30 minutes
  Unexpected immediate adverse events up to 30 minutes post-administration of 18F-fluorocholine.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Probst, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No